CLINICAL TRIAL: NCT05655520
Title: A Phase 3, Multicenter, Open-label Safety Study to Evaluate the Long-term Safety and Tolerability of SAGE-718 in Participants With Huntington's Disease
Brief Title: A Study to Evaluate the Safety and Tolerability of SAGE-718 in Participants With Huntington's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Internal company decision
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 718-CIH-301
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Huntington's Disease
Keywords: Huntington's Disease; SAGE-718
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Direct Rollover) (Experimental): Participants from the studies 718-CIH-201 (NCT05107128) and 718-CIH-202 (NCT05358821) who will sign the informed consent for study 718-CIH-301 ≤7 days after the last day of the corresponding parent study will be enrolled in this cohort. Participants will receive Sage-718, 0.9 milligrams (mg), orally once daily from Day 1 onwards.
  Interventions: Drug: SAGE-718
- Cohort 2 (Gap Rollover) (Experimental): Participants from the studies 718-CIH-201 (NCT05107128) and 718-CIH-202 (NCT05358821) who will sign the informed consent for study 718-CIH-301 after a gap of >7 days after the last day of the corresponding parent study will be enrolled in this cohort. Participants will receive Sage-718 0.9 mg, orally once daily from Day 1 onwards.
  Interventions: Drug: SAGE-718
- Cohort 3 (De Novo) (Experimental): Participants who were not previously included in any SAGE-718 clinical study. Participants will receive Sage-718 from Day 1 onwards.
  Interventions: Drug: SAGE-718

INTERVENTIONS:
Drug: SAGE-718 — Oral softgel lipid capsules

SUMMARY:
The primary purpose of the study is to evaluate the safety and tolerability of SAGE-718 softgel lipid capsule in participants with Huntington's Disease (HD)

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Completed 718-CIH-201 (NCT05107128) or 718-CIH-202 (NCT05358821) studies or meet eligibility criteria for the de novo cohort.
* Agree to refrain from drugs of abuse for the duration of the study and from alcohol during the 48 hours preceding each study visit.
* Be willing to invite a study partner, if available, who is reliable, competent, and at least 18 years of age to participate in the study.
* Be able to travel to the study center, and, judged by the investigator, is likely to be able to continue to travel to the study center to complete study visits for the duration of the study.

Additional inclusion criteria for the de novo cohort (Cohort 3):

* Be at least 25 years old, but not older than 65 years of age at Screening.

  * Genetically confirmed disease with cytosine-adenine-guanine (CAG) expansion ≥40
  * No features of juvenile HD
* CAG-Age-Product (CAP) score ≥90, as calculated using the CAP formula: AGE × (CAG - 30) / 6.49.
* At screening, scores of either: a) Unified Huntington's Disease Rating Scale (UHDRS) -Total Functional Capacity (TFC)=13 and Montreal Cognitive Assessment (MoCA) ≤25 score, or b) UHDRS-TFC ≤12 and MoCA >25

Exclusion Criteria:

For all participants

* Have a diagnosis of an ongoing neurodegenerative condition other than HD, including but not limited to, Alzheimer's Disease, vascular dementia, dementia with Lewy bodies, or Parkinson's Disease.
* Had gastric bypass surgery, has a gastric sleeve or lap band, or has had any related procedures that interfere with gastrointestinal transit.
* Is known to be allergic to any of SAGE-718 excipients, including soy lecithin.
* Receive any prohibited medications within 30 days of screening and during participation in the study.

Additional exclusion criteria for the de novo cohort (Cohort 3):

* Have previous exposure to gene therapy, or have participated in any other HD investigational drug, biologic, or device trial within 180 days or a non-HD drug, biologic or device trial within 30 days or 5 half-lives (whichever is longer). Additionally, participants who have received treatment with antisense oligonucleotides or a messenger ribonucleic acid (mRNA) splicing modifier will be excluded.

Note: Participants with confirmation of enrolment in the placebo arm of these investigational trials would not be excluded.

Additional exclusion criteria for 718-CIH-201/202 completers (Cohorts 1 and 2):

* Have one or more ongoing serious adverse events (SAEs) from the parent study.
* Have ongoing, unresolved AE(s), which in the opinion of the investigator or sponsor, is likely to interfere with study conduct or compliance.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (28):
  - Sage Investigational Site, Birmingham, Alabama
  - Sage Investigational Site, Little Rock, Arkansas
  - Sage Investigational Site, La Jolla, California
  - Sage Investigational Site, Los Alamitos, California
  - Sage Investigational Site, Los Angeles, California
  - Sage Investigational Site, Sacramento, California
  - Sage Investigational Site, Englewood, Colorado
  - Sage Investigational Site, Washington D.C., District of Columbia
  - Sage Investigational Site, Boca Raton, Florida
  - Sage Investigational Site, Tampa, Florida
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Indianapolis, Indiana
  - Sage Investigational Site, Iowa City, Iowa
  - Sage Investigational Site, Kansas City, Kansas
  - Sage Investigational Site, Baltimore, Maryland
  - Sage Investigational Site, Boston, Massachusetts
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Williamsville, New York
  - Sage Investigational Site, Chapel Hill, North Carolina
  - Sage Investigational Site, Durham, North Carolina
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, Toledo, Ohio
  - Sage Investigational Site, Philadelphia, Pennsylvania
  - Sage Investigational Site, Charleston, South Carolina
  - Sage Investigational Site, Memphis, Tennessee
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, Richmond, Virginia
  - Sage Investigational Site, Spokane, Washington
- Australia (3):
  - Sage Investigational Site, Westmead, New South Wales
  - Sage Investigational Site, Caulfield South, Victoria
  - Sage Investigational Site, Nedlands, Western Australia
- Canada (3):
  - Sage Investigational Site, Halifax, Nova Scotia
  - Sage Investigational Site, Toronto, Ontario
  - Sage Investigational Site, Montreal, Quebec
- United Kingdom (8):
  - Sage Investigational Site, Plymouth, Derriford
  - Sage Investigational Site, Southampton, England
  - Sage Investigational Site, Tooting, London
  - Sage Investigational Site, Aberdeen, Scotland
  - Sage Investigational Site, Newcastle, Upon Tyne
  - Sage Investigational Site, Cardiff, Wales
  - Sage Investigational Site, Birmingham, West Midlands
  - Sage Investigational Site, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participation of a study partner was optional in this study and was only to support completion of study activities and answer questions about the participant's condition. Only participants with Huntington's Disease enrolled in this study represented enrollment number. Data presented in all the sections of the results represents data exclusively collected and analyzed for participants with Huntington's Disease enrolled in this study.
Pre-assignment Details: A total of 165 participants were screened, of which, 153 participants were enrolled and received study treatment in either Cohort 1 (Direct rollover) or Cohort 2 (Gap rollover). The study was terminated early by the Sponsor and hence, no participants were enrolled in Cohort 3 (De novo) and therefore no data was collected and reported.
  No additional milestone.
Groups:
- Cohort 1 (Direct Rollover): Participants from the studies 718-CIH-201 (NCT05107128) and 718-CIH-202 (NCT05358821) who signed the informed consent for study 718-CIH-301 ≤7 days after the last day of the corresponding parent study were enrolled in this cohort. Participants received Sage-718, 0.9 milligrams (mg), orally once daily from Day 1 onwards.
- Cohort 2 (Gap Rollover): Participants from the studies 718-CIH-201 (NCT05107128) and 718-CIH-202 (NCT05358821) who signed the informed consent for study 718-CIH-301 after a gap of >7 days following the last day of the corresponding parent study were enrolled in this cohort. Participants received Sage-718, 0.9 mg, orally once daily from Day 1 onwards.
Period: Overall Study
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Started | 72 | 81
Completed | 2 | 4
Not Completed | 70 | 77
Not completed — Adverse Event | 2 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Non-Compliance with Study Drug | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Study Terminated by Sponsor | 61 | 68

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who were administered investigational product (IP) during the study.
Groups:
- Cohort 1 (Direct Rollover): Participants from the studies 718-CIH-201 (NCT05107128) and 718-CIH-202 (NCT05358821) who signed the informed consent for study 718-CIH-301 ≤7 days after the last day of the corresponding parent study were enrolled in this cohort. Participants received Sage-718, 0.9 mg, orally once daily from Day 1 onwards.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover) | Total
Number analyzed (Participants) | 72 | 81 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (8.02) | 51.2 (9.21) | 51.6 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 38 | 72
  Male | 38 | 43 | 81
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 1 | 0 | 1
  Race: Black or African American | 0 | 2 | 2
  Race: Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Race: White | 68 | 77 | 145
  Race: Multiple | 0 | 1 | 1
  Race: Other | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanice or Latino | 8 | 5 | 13
  Ethnicity: Not Hispanic or Latino | 64 | 76 | 140

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE is defined as an AE with onset after the start of IP, or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study.
Time Frame: Up to 24 months
Population: The Safety Set included all participants who were administered IP during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 72 | 81
Participants | 46 | 46

2. Primary Outcome: Number of Participants With at Least One TEAE by Severity
Description: A TEAE is defined as an AE with onset after the start of IP, or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study. Severity was assessed as:
  Mild: symptoms barely noticeable to participant or does not make participant uncomfortable; does not influence performance or functioning; prescription drug not ordinarily needed for relief of symptoms.
  Moderate: symptoms of a sufficient severity to make participant uncomfortable; performance of daily activity is influenced; participant is able to continue in study; treatment for symptoms may be needed.
  Severe: symptoms cause severe discomfort; symptoms cause incapacitation or significant impact on participant's daily life; severity may cause cessation of treatment with IP; treatment for symptoms may be given and/or participant hospitalized.
  Participant with multiple instances of events is counted only once using maximum intensity.
Time Frame: Up to 24 months
Population: The Safety Set included all participants who were administered IP during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 72 | 81
Participants
  Mild | 21 | 24
  Moderate | 22 | 18
  Severe | 3 | 4

3. Primary Outcome: Number of Participants Who Withdrew From Study Due to TEAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE is defined as any AE with onset or after the start of IP or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study.
Time Frame: Up to 24 months
Population: The Safety Set included all participants who were administered IP during the study.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 (Direct Rollover): Participants from the studies 718-CIH-201 (NCT05107128) and 718-CIH-202 (NCT05358821) who signed the informed consent for study 718-CIH-301 ≤7 days after the last day of the corresponding parent study were enrolled in this cohort. Participants received Sage-718 0.9 mg, orally once daily from Day 1 onwards.
- Cohort 2 (Gap Rollover): Participants from the studies 718-CIH-201 (NCT05107128) and 718-CIH-202 (NCT05358821) who signed the informed consent for study 718-CIH-301 after a gap of >7 days after the last day of the corresponding parent study were enrolled in this cohort. Participants received Sage-718, 0.9 mg, orally once daily from Day 1.
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 72 | 81
Participants | 2 | 3

4. Primary Outcome: Change From Baseline in Vital Signs: Blood Pressure
Description: Vital signs parameter for blood pressure included systolic blood pressure (supine), systolic blood pressure (standing 1 minute), systolic blood pressure (standing 3 minutes), diastolic blood pressure (supine), diastolic blood pressure (standing 1 minute), and diastolic blood pressure (standing 3 minutes).
  Last value on study is defined as the last post-baseline value on or after the first dose of IP and on or before the last date of the study.
Time Frame: Baseline; Last Value on Study (up to 24 months)
Population: The Safety Set included all participants who were administered IP during the study. Overall number of participants analyzed are the participants who were evaluable for vital sign parameters for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 71 | 80
mmHg
  Change From Baseline (CFB): Systolic Blood Pressure (Supine) | 0.2 (11.49) | 0.4 (14.61)
  CFB: Systolic Blood Pressure (Standing 1 minute) | -1.8 (17.63) | 1.0 (14.72)
  CFB: Systolic Blood Pressure (Standing 3 minute) | -2.0 (13.85) | -0.3 (13.94)
  CFB: Diastolic Blood Pressure (Supine) | 1.2 (8.10) | -1.1 (9.02)
  CFB: Diastolic Blood Pressure (Standing 1 minute) | 1.4 (11.41) | -0.7 (10.27)
  CFB: Diastolic Blood Pressure (Standing 3 minute) | 0.5 (10.33) | -1.3 (11.02)

5. Primary Outcome: Change From Baseline in Vital Signs: Heart Rate
Description: Vital signs for heart rate included heart rate (supine), heart rate (standing 1 minute), and heart rate (standing 3 minute).
  Last value on study is defined as the last post-baseline value on or after the first dose of IP and on or before the last date of the study.
Time Frame: Baseline, Last value on study (up to 24 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 71 | 80
beats/min
  CFB: Heart Rate Supine | 2.2 (9.66) | 2.7 (9.91)
  CFB: Heart Rate Standing 1 Minute | 1.8 (13.13) | 2.2 (11.45)
  CFB: Heart Rate Standing 3 Minute | 1.7 (12.65) | 2.1 (14.00)

6. Primary Outcome: Change From Baseline in Vital Signs: Respiratory Rate
Description: Last value on study is defined as the last post-baseline value on or after the first dose of IP and on or before the last date of the study.
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 71 | 80
breaths/min | 0.0 (2.64) | -0.1 (2.76)

7. Primary Outcome: Change From Baseline in Vital Signs: Temperature
Description: as for outcome 6
Time Frame: Baseline, Last value on study (up to 24 months)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 71 | 80
degree Celsius | 0.9 (7.519) | 0.058 (0.3650)

8. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Hematology - Basophils, Eosinophils, Erythrocytes, Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: The Safety Set included all participants who were administered IP during the study. Overall number of participants analyzed are the participants who were evaluable for clinical laboratory parameters for this outcome measure and Number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 68 | 78
cells*10^9/L
  CFB: Basophils | 0.00 (0.039) | 0.01 (0.052)
  CFB: Eosinophils | 0.00 (0.091) | 0.02 (0.101)
  CFB: Erythrocytes | 0.004 (0.2369) | 0.015 (0.2312)
  CFB: Leukocytes | -0.21 (1.609) | 0.07 (1.328)
  CFB: Lymphocytes | -0.03 (0.317) | -0.04 (0.362)
  CFB: Monocytes | 0.01 (0.134) | 0.03 (0.115)
  CFB: Neutrophils | -0.20 (1.561) | 0.06 (1.230)
  CFB: Platelets: number analyzed (Participants) | 68 | 77
  CFB: Platelets | 6.6 (37.38) | 4.2 (30.31)

9. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Hematology- Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes, Neutrophils/Leukocytes
Description: as for outcome 6
Time Frame: Baseline, Last value on study (up to 24 months)
Population: The Safety Set included all participants who were administered IP during the study. Overall number of participants analyzed are the participants who were evaluable for clinical laboratory parameters for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 68 | 78
percent
  CFB: Basophils/Leukocytes | 0.02 (0.313) | -0.02 (0.240)
  CFB: Eosinophils/Leukocytes | 0.04 (1.259) | 0.32 (1.268)
  CFB: Lymphocytes/Leukocytes | -0.11 (6.984) | -0.66 (6.023)
  CFB: Monocytes/Leukocytes | 0.32 (2.427) | 0.57 (1.547)
  CFB: Neutrophils/Leukocytes | -0.25 (8.792) | -0.20 (7.208)

10. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Hematology- Erythrocytes (Ery.) Mean Corpuscular Hemoglobin (HGB) Concentration, Hemoglobin
Description: as for outcome 6
Time Frame: Baseline, Last value on study (up to 24 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 68 | 78
grams per liter (g/L)
  CFB: Ery. Mean Corpuscular HGB Concentration | -2.7 (11.85) | -4.9 (9.24)
  CFB: Hemoglobin | -0.0 (6.69) | -0.3 (8.15)

11. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Hematology - Erythrocytes Mean Corpuscular Hemoglobin
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 68 | 78
picograms (pg) | -0.02 (0.740) | -0.17 (0.953)

12. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Hematology - Erythrocytes Mean Corpuscular Volume
Description: as for outcome 6
Time Frame: Baseline, Last value on study (up to 24 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: femtoliters (fL)
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 68 | 78
femtoliters (fL) | 0.61 (3.091) | 0.85 (2.884)

13. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Hematology - Hematocrit
Description: as for outcome 6
Time Frame: Baseline, Last value on study (up to 24 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: liters per liter (L/L)
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 68 | 78
liters per liter (L/L) | 0.0033 (0.0256) | 0.0055 (0.0271)

14. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Biochemistry- Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Creatine Kinase, Gamma Glutamyl Transferase, Lactate Dehydrogenase
Description: as for outcome 6
Time Frame: Baseline, Last value on study (up to 24 months)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 71 | 79
units per liter (U/L)
  CFB: Alanine Aminotransferase: number analyzed (Participants) | 68 | 79
  CFB: Alanine Aminotransferase | -1.2 (10.80) | 0.6 (11.42)
  CFB: Alkaline Phosphatase | 1.7 (13.17) | 2.2 (13.04)
  CFB: Aspartate Aminotransferase: number analyzed (Participants) | 68 | 79
  CFB: Aspartate Aminotransferase | -1.7 (5.56) | 1.0 (9.79)
  CFB: Creatinine Kinase | -28.6 (135.53) | -0.8 (83.46)
  CFB: Gamma Glutamyl Transferase | 3.1 (14.47) | 4.0 (31.75)
  CFB: Lactate Dehydrogenase: number analyzed (Participants) | 67 | 78
  CFB: Lactate Dehydrogenase | -9.6 (19.89) | 4.2 (25.26)

15. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Biochemistry - Bicarbonate, Calcium, Chloride, Cholesterol, Glucose, HDL Cholesterol, LDL Cholesterol, Phosphate, Potassium, Sodium, Triglycerides, Urea Nitrogen
Description: HDL= high-density lipoprotein LDL= low-density lipoprotein
  Last value on study is defined as the last post-baseline value on or after the first dose of IP and on or before the last date of the study.
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 71 | 79
millimole per liter (mmol/L)
  CFB: Bicarbonate: number analyzed (Participants) | 71 | 78
  CFB: Bicarbonate | -0.1 (2.68) | 0.0 (2.51)
  CFB: Calcium: number analyzed (Participants) | 70 | 79
  CFB: Calcium | -0.005 (0.0905) | 0.006 (0.0861)
  CFB: Chloride: number analyzed (Participants) | 70 | 79
  CFB: Chloride | 0.7 (2.31) | 1.0 (2.31)
  CFB: Cholesterol | -0.02 (0.777) | 0.22 (0.735)
  CFB: Glucose: number analyzed (Participants) | 67 | 78
  CFB: Glucose | -0.04 (1.128) | -0.26 (1.274)
  CFB: HDL Cholesterol | -0.00 (0.188) | 0.05 (0.218)
  CFB: LDL Cholesterol | -0.01 (0.636) | 0.08 (0.671)
  CFB: Phosphate: number analyzed (Participants) | 68 | 78
  CFB: Phosphate | 0.009 (0.1688) | -0.017 (0.1937)
  CFB: Potassium: number analyzed (Participants) | 67 | 78
  CFB: Potassium | -0.07 (0.463) | -0.06 (0.319)
  CFB: Sodium: number analyzed (Participants) | 70 | 79
  CFB: Sodium | 0.4 (1.99) | 0.7 (2.02)
  CFB: Triglycerides | -0.125 (0.9411) | 0.080 (0.8615)
  CFB: Urea Nitrogen | 0.33 (1.371) | -0.11 (1.344)

16. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Biochemistry - Albumin and Protein
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 71 | 79
grams per liter (g/L)
  CFB: Albumin | 0.2 (2.78) | 0.4 (2.11)
  CFB: Protein | -1.0 (3.60) | -0.2 (3.09)

17. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Biochemistry - Bilirubin, Creatinine, Direct Bilirubin, Indirect Bilirubin
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: micromoles per liter (µmol/L)
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 71 | 79
micromoles per liter (µmol/L)
  CFB: Bilirubin | -0.43 (3.149) | -0.10 (2.912)
  CFB: Creatinine | 0.7 (8.14) | 3.0 (9.95)
  CFB: Direct Bilirubin | -0.04 (1.201) | -0.25 (1.223)
  CFB: Indirect Bilirubin | -0.39 (2.367) | 0.15 (2.137)

18. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Biochemistry - Thyrotropin
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milli-international units per liter
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 71 | 79
milli-international units per liter | -0.061 (2.2278) | -0.181 (1.2943)

19. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Biochemistry - Thyroxine Free, Triiodothyronine Free
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: picomoles per liter (pmol/L)
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 2 | 1
picomoles per liter (pmol/L)
  CFB: Thyroxine, Free | 2.55 (20.153) | 6.40 (NA) — Standard deviation could not be calculated due to low number of participants available for analysis.
  CFB: Triiodothyronine, Free | 0.85 (1.909) | 1.70 (NA) — Standard deviation could not be calculated due to low number of participants available for analysis.

20. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Urinalysis- Erythrocytes in Urine, Leukocytes in Urine, Renal Epithelial Casts, Squamous Epithelial Cells, Transitional Epithelial Cells
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cells per high power field
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 11 | 19
cells per high power field
  CFB: Erythrocytes in Urine | 0.9 (3.30) | -0.2 (2.09)
  CFB: Leukocytes in Urine: number analyzed (Participants) | 10 | 19
  CFB: Leukocytes in Urine | -2.4 (4.45) | 0.8 (7.53)
  CFB: Renal Epithelial Casts | 0.00 (0.00) | 0.00 (0.00)
  CFB: Squamous Epithelial Cells | -1.3 (16.29) | 0.8 (4.98)
  CFB: Transitional Epithelial Cells | 0.0 (0.89) | 0.5 (1.12)

21. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Urinalysis- Hyaline Casts
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: casts per low power field (/lpf)
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 11 | 19
casts per low power field (/lpf) | 0.9 (3.56) | -0.6 (1.89)

22. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Urinalysis- pH
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 68 | 78
pH | -0.13 (0.667) | 0.06 (0.679)

23. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Coagulation- Activated Partial Thromboplastin Time, Prothrombin Time
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 68 | 80
seconds
  CFB: Activated Partial Thromboplastin Time | 0.86 (5.876) | -1.12 (2.947)
  CFB: Prothrombin Time | 0.14 (1.008) | -0.05 (0.673)

24. Primary Outcome: Change From Baseline in Clinical Laboratory Parameters: Coagulation- Prothrombin International (Intl) Normalized Ratio
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: prothrombin intl normalized ratio
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 68 | 80
prothrombin intl normalized ratio | 0.011 (0.1071) | -0.011 (0.0740)

25. Primary Outcome: Change From Baseline in Electrocardiograms (ECGs) Parameters: Mean Heart Rate
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: The Safety Set included all participants who were administered IP during the study. Overall number of participants analyzed are the participants who were evaluable for ECG parameter for this outcome measure.
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 68 | 80
beats per minute (beats/min) | 1.3 (9.54) | 1.6 (8.80)

26. Primary Outcome: Change From Baseline in ECG Parameters - PR Interval Aggregate, QRS Duration Aggregate, QT Interval Aggregate and QTcF Interval Aggregate
Description: as for outcome 6
Time Frame: Baseline; Last value on study (up to 24 months)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 68 | 80
millisecond (msec)
  CFB: PR Interval, Aggregate | -2.8 (13.39) | -0.2 (12.94)
  CFB: QRS Duration, Aggregate | 1.8 (9.0) | -0.8 (9.11)
  CFB: QT Interval, Aggregate | -1.4 (22.72) | -2.9 (20.94)
  CFB: QTcF Interval, Aggregate | 0.8 (15.32) | -0.0 (14.81)

27. Primary Outcome: Number of Participants With Change From Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) Responses
Description: Columbia Suicide Severity Rating Scale evaluates and assesses the lifetime experience of participants with suicidal ideation (SI) and suicidal behavior (SB) and post-baseline evaluation that focuses on suicidality since last study visit. C-SSRS includes "yes" or "no"' responses for assessment of SI and SB as well as numeric ratings for severity of ideation. If present [from 1 (minor physical damage) to 5 (death), with 5 being most severe]. If any of the available assessments in suicidal behavior is Yes, the category is considered as 'Suicidal behavior'. If any of these available assessments in suicidal ideation is Yes but all available assessments in suicidal behavior is NO, the category is considered as 'Suicidal Ideation'. Data is reported for only those timepoints where there was a change in assessment (response) from Baseline. Baseline is the worst of assessments done in any question in SI/SB prior to first dose of IP, excluding lifetime assessment.
Time Frame: Day 30, Day 60, Day 90, Day 365, Day 395, Safety Follow-up (up to 24 months)
Population: The Safety Set included all participants who were administered IP during the study. Number analyzed is the number of participants with data available for analysis at specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
Number analyzed (Participants) | 72 | 81
Participants
  Day 30: number analyzed (Participants) | 65 | 74
  Day 30: No suicidal ideation/behavior to No suicidal ideation/behavior | 65 | 73
  Day 30: No suicidal ideation/behavior to Suicidal ideation | 0 | 0
  Day 30: No suicidal ideation/behavior to Suicidal Behavior | 0 | 0
  Day 30: Suicidal Ideation to No suicidal ideation/behavior | 0 | 1
  Day 30: Suicidal Ideation to Suicidal Ideation | 0 | 0
  Day 30: Suicidal Ideation to Suicidal Behavior | 0 | 0
  Day 30: Suicidal Behavior to No suicidal ideation/behavior | 0 | 0
  Day 30: Suicidal Behavior to Suicidal Ideation | 0 | 0
  Day 30: Suicidal Behavior to Suicidal Behavior | 0 | 0
  Day 60: number analyzed (Participants) | 60 | 70
  Day 60: No suicidal ideation/behavior to No suicidal ideation/behavior | 59 | 69
  Day 60: No suicidal ideation/behavior to Suicidal ideation | 1 | 0
  Day 60: No suicidal ideation/behavior to Suicidal Behavior | 0 | 0
  Day 60: Suicidal Ideation to No suicidal ideation/behavior | 0 | 1
  Day 60: Suicidal Ideation to Suicidal Ideation | 0 | 0
  Day 60: Suicidal Ideation to Suicidal Behavior | 0 | 0
  Day 60: Suicidal Behavior to No suicidal ideation/behavior | 0 | 0
  Day 60: Suicidal Behavior to Suicidal Ideation | 0 | 0
  Day 60: Suicidal Behavior to Suicidal Behavior | 0 | 0
  Day 90: number analyzed (Participants) | 53 | 64
  Day 90: No suicidal ideation/behavior to No suicidal ideation/behavior | 51 | 63
  Day 90: No suicidal ideation/behavior to Suicidal ideation | 2 | 0
  Day 90: No suicidal ideation/behavior to Suicidal Behavior | 0 | 0
  Day 90: Suicidal Ideation to No suicidal ideation/behavior | 0 | 1
  Day 90: Suicidal Ideation to Suicidal Ideation | 0 | 0
  Day 90: Suicidal Ideation to Suicidal Behavior | 0 | 0
  Day 90: Suicidal Behavior to No suicidal ideation/behavior | 0 | 0
  Day 90: Suicidal Behavior to Suicidal Ideation | 0 | 0
  Day 90: Suicidal Behavior to Suicidal Behavior | 0 | 0
  Day 365: number analyzed (Participants) | 20 | 32
  Day 365: No suicidal ideation/behavior to No suicidal ideation/behavior | 20 | 31
  Day 365: No suicidal ideation/behavior to Suicidal ideation | 0 | 0
  Day 365: No suicidal ideation/behavior to Suicidal Behavior | 0 | 0
  Day 365: Suicidal Ideation to No suicidal ideation/behavior | 0 | 0
  Day 365: Suicidal Ideation to Suicidal Ideation | 0 | 0
  Day 365: Suicidal Ideation to Suicidal Behavior | 0 | 1
  Day 365: Suicidal Behavior to No suicidal ideation/behavior | 0 | 0
  Day 365: Suicidal Behavior to Suicidal Ideation | 0 | 0
  Day 365: Suicidal Behavior to Suicidal Behavior | 0 | 0
  Day 395: number analyzed (Participants) | 7 | 8
  Day 395: No suicidal ideation/behavior to No suicidal ideation/behavior | 7 | 7
  Day 395: No suicidal ideation/behavior to Suicidal ideation | 0 | 0
  Day 395: No suicidal ideation/behavior to Suicidal Behavior | 0 | 0
  Day 395: Suicidal Ideation to No suicidal ideation/behavior | 0 | 0
  Day 395: Suicidal Ideation to Suicidal Ideation | 0 | 1
  Day 395: Suicidal Ideation to Suicidal Behavior | 0 | 0
  Day 395: Suicidal Behavior to No suicidal ideation/behavior | 0 | 0
  Day 395: Suicidal Behavior to Suicidal Ideation | 0 | 0
  Day 395: Suicidal Behavior to Suicidal Behavior | 0 | 0
  Safety Follow-up (up to 24 months): number analyzed (Participants) | 50 | 59
  Safety Follow-up (up to 24 months): No suicidal ideation/behavior to No suicidal ideation/behavior | 50 | 58
  Safety Follow-up (up to 24 months): No suicidal ideation/behavior to Suicidal ideation | 0 | 0
  Safety Follow-up (up to 24 months): No suicidal ideation/behavior to Suicidal Behavior | 0 | 0
  Safety Follow-up (up to 24 months): Suicidal Ideation to No suicidal ideation/behavior | 0 | 1
  Safety Follow-up (up to 24 months): Suicidal Ideation to Suicidal Ideation | 0 | 0
  Safety Follow-up (up to 24 months): Suicidal Ideation to Suicidal Behavior | 0 | 0
  Safety Follow-up (up to 24 months): Suicidal Behavior to No suicidal ideation/behavior | 0 | 0
  Safety Follow-up (up to 24 months): Suicidal Behavior to Suicidal Ideation | 0 | 0
  Safety Follow-up (up to 24 months): Suicidal Behavior to Suicidal Behavior | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: The Safety Set included all participants who were administered IP during the study.
Arm/Group | Cohort 1 (Direct Rollover) | Cohort 2 (Gap Rollover)
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/81
Serious Adverse Events (participants affected / at risk) | 3/72 | 6/81
Other Adverse Events (participants affected / at risk) | 46/72 | 22/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Direct Rollover) (N=72) | Cohort 2 (Gap Rollover) (N=81)
Psychotic disorder (Psychiatric disorders) | 1 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Huntington's disease (Congenital, familial and genetic disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Direct Rollover) (N=72) | Cohort 2 (Gap Rollover) (N=81)
Fall (Injury, poisoning and procedural complications) | 6 | 9
Nasopharyngitis (Infections and infestations) | 6 | 4
Depression (Psychiatric disorders) | 5 | 4
Anxiety (Psychiatric disorders) | 5 | 2
Balance disorder (Nervous system disorders) | 4 | 3
Chorea (Nervous system disorders) | 4 | 3
Insomnia (Psychiatric disorders) | 4 | 3
Contusion (Injury, poisoning and procedural complications) | 4 | 2
Gait disturbance (General disorders) | 4 | 2
Skin laceration (Injury, poisoning and procedural complications) | 4 | 2
Somnolence (Nervous system disorders) | 5 | 1
Suicidal ideation (Psychiatric disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT05655520/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT05655520/SAP_001.pdf